CLINICAL TRIAL: NCT04593368
Title: Prospective Non-randomized Phase II Clinical Trial of Safety and Efficacy of Fecal Microbiome Transplantation for Pediatric Patients 3-18 Years Old With Confirmed Colonization With Antibiotic-resistant Bacterias and Indication for Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Fecal Microbiome Transplantation (FMT) in Pediatric Patients Colonized With Antibiotic-resistant Pathogens Before Hematopoietic Stem Cell Transplantation (HSCT)
Acronym: FMT-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCPHOI-2019-04
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Antibiotic Resistant Strain
Keywords: pediatric; hematopoetic stem-cell transplantation; FMT; microbiome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental)
  Interventions: Other: FMT

INTERVENTIONS:
Other: FMT — oral dosing of fecal microbiome from allogeneic donor, 0.5-2 g/kg of recipients weight

SUMMARY:
a clinical trial designed to prospectively assess the safety and effectiveness of fecal microbiota transplantation (FMT) prior to allogeneic hematopoietic stem-cell translation (HSCT) in patients contaminated with antibiotic-resistant pathogens (ARP)

DETAILED DESCRIPTION:
The investigator's question is whether FMT decontaminates ARP and as a result, decreases the risk of severe infection which leads to transplant-related morbidity and mortality after HSCT.

ELIGIBILITY:
Recipients

Inclusion Criteria:

1. detection by microbiology culture in any localization species of:

   * Pseudomonas aeruginosa
   * Clostridium difficile
   * Vancomycin-resistant Enterococcus
   * Streptococcus viridans
   * ESBL Enterobacteriaceae, including Escherichia coli and Klebsiella pneumoniae
   * Stenotrophomonas maltophilia
   * Acinetobacter
   * Methicillin-resistant Staphylococcus aureus
2. Indications for allo-HSCT

Exclusion Criteria:

1. indications for therapy with antibiotics for the next 7 days after FMT
2. Nonstable condition during 1 week before FMT
3. Therapy with antibiotics less than 48 hours before FMT
4. Age less than 3 years
5. Neutrophils count < 0,5 K/mcL at FMT day and\or predicted decrease during 2 days after Donors (healthy volunteers)

Inclusion Criteria:

1. Age 3-50 years old
2. Donor choosing order in the absence of contraindications:

1) HLA-match/mismatch HSCT family donor; 2) Closest family relative with whom the recipient lives; 3) Unrelated healthy volunteer from the FRCC PCM bank of frozen transplants

Exclusion Criteria:

1. Presens of:

   * ESBL Esherihia coli
   * Klebsiella pneumoniae
   * Pseudomonas aeruginosa
   * Clostridium difficile
   * MRSA
   * VRE
   * Streptococcus viridans
   * ESBL Enterobacteriaceae
   * Stenotrophomonas maltophilia
   * Acinetobacter in feces by microbiology culture assay
2. Therapy with antibiotics less than 3 months before donation
3. Any infection disease revealed during the screening
4. Latent period of infection disease according to the questionnaire
5. Gut disease
6. Longitudinal treatment with drugs
7. Any diet for 3 months before donation.
8. Obesity (BMI ≥ 30).

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 7 days after FMT
  frequency of decolonization
frequency of SAEs | 1 month after FMT
  frequency of SAEs due to FMT

SECONDARY OUTCOMES:
Decolonization | 30 days after FMT
  frequency of decolonization
acute gut GVHD CI | 100 days after HSCT
  CI of gut GVHD
Toxicity frequency | 7 days after FMT
  frequency of severe toxicity (3-4 grade according to the CTCAE ver 5.0)
Bacteremia | 100 days after FMT
  frequency of bacteremia
Translocation | 1 year
  frequency of translocation of pathogens from gut

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow
  - Federal Research & Clinical Center of Physical-Chemical Medicine of Federal Medical Biological Agency, Moscow
  - RM Gorbacheva Research Institute of Pediatric Oncology, Hematology and Transplantation, Pavlov University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No